CLINICAL TRIAL: NCT04939805
Title: Selective C-reactive Protein Apheresis in ST-elevation Myocardial Infarction
Brief Title: CRP Apheresis in STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210121-2475
Record Dates: First submitted 2021-06-07; First posted 2021-06-25 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: ST Elevation Myocardial Infarction; C-Reactive Protein; Apheresis; Myocardial Injury
Keywords: Cardiac magnetic resonance imaging
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective CRP apheresis as an adjunct to standard of care (Experimental): Apheresis using the PentraSorb®-CRP system will be performed at day 1, 2 and 3 after PCI.
  Interventions: Device: Selective CRP apheresis using the PentraSorb®-CRP system
- Standard of care according to current guideline recommendations (No Intervention)

INTERVENTIONS:
Device: Selective CRP apheresis using the PentraSorb®-CRP system — Selective CRP apheresis as an adjunct to standard of care. Apheresis using the PentraSorb®-CRP system will be performed at day 1, 2 and 3 after PCI.
  Arms: Selective CRP apheresis as an adjunct to standard of care

SUMMARY:
Background: In patients with acute ST-elevation myocardial infarction (STEMI), the amount of infarcted myocardium (infarct size) is known to be a major predictor for adverse remodeling and recurrent adverse cardiovascular events. Effective cardio-protective strategies with the aim of reducing infarct size are therefore of great interest. Local and systemic inflammation influences the fate of ischemic myocardium and thus, adverse remodeling and clinical outcome. C-reactive protein (CRP) also acts as a potential mechanistic mediator that adversely affects the amount of irreversible myocardial tissue damage after acute myocardial infarction.

Objective: The main objectives of the current study are to investigate the efficacy of selective CRP apheresis, using the PentraSorb®-CRP system, as an adjunctive therapy to standard of care for patients with acute STEMI treated with primary PCI.

Design: Investigator-initiated, prospective, randomized, open-label (outcome assessors masked), controlled, multicenter, two group trial with a two-stage adaptive design.

Innovation: Selective CRP apheresis offers potential to decrease infarct size and consequently improve outcome after PCI for STEMI. This is the first randomized trial investigating the impact of selective CRP apheresis on infarct size in post-STEMI patients. In perspective, the study design allows furthermore to collect robust evidence for the design of a definitive outcome study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of first acute STEMI in accordance with the European Society of Cardiology (ESC) Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation
2. Symptoms consistent with STEMI with beginning greater than 30 minutes but less than 12 hours prior to primary percutaneous coronary intervention (PCI)
3. CRP elevation of ≥7 mg/l measured between 6 to 16 hours after primary PCI
4. Eligible for primary PCI
5. Age ≥18 years
6. Written informed consent

Exclusion Criteria:

1. Prior acute myocardial infarction, coronary artery bypass surgery or PCI.
2. Persistent hemodynamic instability (Killip class >2 including cardiogenic shock) or resuscitated cardiac arrest not allowing a CMR scan.
3. The patient is febrile (temperature >38°C) or has experienced an acute infection with fever in the last 14 days.
4. CRP >15 mg/l at time of hospital admission.
5. Chronic inflammatory disease.
6. Known history of severe hepatic failure
7. Chronic kidney disease with a creatinine clearance <30ml/min./1.73m²
8. Contraindication to CMR.
9. Pre-STEMI life expectancy of <1 year
10. Participation in another interventional trial
11. Limited possibility to join the follow-up examinations (e.g. patient lives abroad)
12. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 5 ± 2 days post PCI
  Infarct size expressed as % of left ventricular myocardial mass (LVMM) as visualized by cardiac magnetic resonance (CMR) imaging at 5 ± 2 days post PCI

SECONDARY OUTCOMES:
Safety endpoint | during hospitalization for the index event
  Adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) during hospitalization for the index event
All-cause mortality or hospitalization for heart failure within 12 months after randomization | within 12 months after randomization
  All-cause mortality or hospitalization for heart failure within 12 months after randomization (endpoint of interest with respect to the two-stage adaptive design)
CMR endpoints defined as: Left ventricular ejection fraction and microvascular obstruction and exploratory (intramyocardial hemorrhage, edema extent, myocardial salvage, native T1 mapping, strain) | at baseline, 4 months and 12 months after PCI for STEMI
  CMR endpoints will be assessed at baseline, 4 and 12 months CMR follow-up study and are defined according to the Journal of American College of Cardiology Scientific Expert Consensus document.
Hospitalization for heart failure within 12 months after randomization | within 12 months after randomization
Cardiovascular mortality at 12 months | within 12 months after randomization
CRP concentrations | during hospitalization for the index event
  CRP concentrations during index hospitalization
Left ventricular thrombus formation | 5 ± 2 days, 4 months, 12 months post PCI
Biomarker concentrations of myocardial necrosis (enzymatic infarct size; high-sensitivity troponin T) | at baseline, 4 months, 12 months post PCI
Biomarker concentrations of hemodynamic stress (N-terminal pro-B-Type Natriuretic Peptide) | at baseline, 4 months, 12 months post PCI
Renal function (eGFR) | during hospitalization for the index event
  as measured by the MDRD and CKD-EPI formula
Renal function (Cystatin C-based calculation of creatinine clearance) | during hospitalization for the index event
Cardiac autonomic function: Deceleration capacity of heart rate | 5 ± 2 days, 4 months, 12 months post PCI
Cardiac autonomic function: Heart rate variability | 5 ± 2 days, 4 months, 12 months post PCI
Cardiac autonomic function: Periodic repolarization dynamics | 5 ± 2 days, 4 months, 12 months post PCI
Cardiac autonomic function: Baroreflex sensitivity | 5 ± 2 days, 4 months, 12 months post PCI
Cardiac autonomic function: Skin sympathetic nerve activity | 5 ± 2 days, 4 months, 12 months post PCI

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian J Reinstadler, MD, PhD, Principal Investigator — University Clinic of Internal Medicine III, Cardiology and Angiology, Medical University of Innsbruck
Locations (5):
- Austria (3):
  - University Clinic for Cardiology and Nephrology, Medical University of Graz, Graz
  - University Clinic of Internal Medicine III, Cardiology and Angiology. University Clinic of Internal Medicine IV, Nephrology and Hypertensiology. University Clinic of Radiology., Innsbruck
  - University Clinic of Internal Medicine II, Paracelsus Medical University Salzburg, Salzburg
- Germany (2):
  - Medical Clinic II - University Heart Center Lübeck, Lübeck, Schleswig-Holstein
  - Leipzig Heart Center, Leipzig

REFERENCES:
- [Derived] Reinstadler SJ, Kronbichler A, Reindl M, Tiller C, Holzknecht M, Oberhollenzer F, Kaser A, Gauckler P, Stiermaier T, Feistritzer HJ, Mayr A, Gizewski ER, Rezar R, Bugger H, Eller K, Eitel I, Schneider S, Mayer G, Thiele H, Bauer A, Metzler B, Lechner I; CRP-STEMI Investigators. Selective C-reactive protein apheresis in ST-elevation myocardial infarction: Design and rationale of the randomized CRP-STEMI trial. Am Heart J. 2026 Jan;291:1-9. doi: 10.1016/j.ahj.2025.07.067. Epub 2025 Jul 28. PMID 40738310